CLINICAL TRIAL: NCT06820684
Title: Inflammatory Response to OMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Northwest University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-05
Record Dates: First submitted 2025-01-16; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Inflammation; Inflammatory Response
MeSH Terms: conditions — Inflammation | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: One group, single-center, non-randomized, pilot evaluation of a one-time brief (10-min) intervention of osteopathic manipulative treatment (OMT) intervention to measure effects on inflammation (TNF-α, IL-6, IL-1β, and IL-10) in healthy adult volunteers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osteopathic Manipulative Treatment (OMT) (Experimental): There will be only one arm for this study. All participants will receive the OMT intervention.
  Interventions: Procedure: Osteopathic Manipulative Treatment (OMT)

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment (OMT) — The OMT protocol will be delivered as follows:
  1. Touching and applying gentle pressure to the participant's upper shoulder area (this is called Thoracic inlet direct myofascial release)
  2. Touching and applying gentle pressure to the participant's midsection and abdomen (this is called Abdominal diaphragm direct myofascial release)
  3. Touching and applying gentle pressure to the participant's pelvis and sacrum (this is called Muscle Energy or Counterstrain, if indicated).
  4. Touching and applying gentle pressure to the participant's hips and hamstrings (this is called muscle energy) and will be done in 3 repeated rounds of 5 seconds each.
  5. Touching and applying gentle pressure to the backs of the participant's knees (this is called open popliteal fossa with direct myofascial release)
  6. Touching and applying gentle pressure to the participant's feet, moving them back and forth in 10 rhythmic pulses (this is called Pedal Pump)

SUMMARY:
Investigators will evaluate inflammation before and after an osteopathic manipulative treatment (OMT) in healthy adults, 18-59 years of age. Investigators will look at proteins in the blood called "cytokines". Cytokines can be pro-inflammatory, or anti-inflammatory. Investigators think OMT will reduce pro-inflammatory cytokines and increase anti-inflammatory cytokines. Investigators have selected 4 cytokines (out of a potential 30) that investigators believe, based on the literature, are most likely to change over a brief time period. This project will lay essential groundwork at the investigators' institution for future research where they will study the effects of OMT in persons with diabetes (DM) and diabetic peripheral neuropathy (DPN). DPN is a common complication of DM and has few treatment options. OMT has never been specifically studied as a treatment for DPN, and if this pilot study shows significant findings, future work in adults with DPN could be useful.

If investigators detect no changes in cytokines, this pilot work is still important. Investigators need to confirm selected tests are sensitive enough to pick up baseline levels of cytokines in healthy people, where there is expected to be low levels of pro-inflammatory markers (IL-6, TNF-alpha, IL-1b), and higher levels of anti-inflammatory markers (IL-10). Investigators will also use these data as comparison for future work in people with expectedly higher levels of inflammation due to diabetes with complications (e.g., DPN). If markers measured in this pilot study don't show anything, investigators can look at additional cytokines in future analyses. Lastly, it's clear that most people have chronic low-level inflammation without showing or experiencing overt disease; there is a likelihood that investigators will still detect changes, even in a healthy population.

DETAILED DESCRIPTION:
Study Hypothesis:

1. OMT will reduce acute pro-inflammatory markers.
2. OMT will increase acute anti-inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* At least 110 lbs.
* Age within stated required range of 18-59 years of age
* BMI <35
* Non-pregnant
* Generally healthy by self-report
* Free from chronic conditions
* Not taking any daily medications
* Willing to abstain from substance use including alcohol and tobacco for 48 hours prior to blood collection
* Willing to fast for 8 hours before blood draw
* Willing to refrain from exercising >48-hr prior to the study visit
* Willing to abstain from abstain from anti-inflammatory medications (e.g., NSAIDs) for at least one week prior to the study visit
* Free of cold and flu symptoms the day of collection
* No infections within two weeks prior to collection
* No symptoms of a heart condition within the six months prior to collection
* No known blood disorder or blood clotting disorder
* No known sickle cell disease
* No known anemia
* Including the study draw, blood donation for clinical or research purposes during the preceding eight weeks will not exceed 550 ml
* No more than one blood draw has occurred during the preceding week

Exclusion Criteria:

* Not in the required age range
* Use of daily medications
* Unable or unwilling to meet the inclusion criteria
* Additional diagnostic tests or urgent/emergent procedures needed beyond study exam procedures
* Any history of vertebral artery pathology
* Any history of congestive heart failure
* Any history of diagnosed or suspected osteoporosis
* Any recent (90 days) infections, inflammatory condition, fractures, surgery, anesthesia, or traumas
* History of malignancies, autoimmune disease, radiation, or chemotherapy at any time
* Individuals with severe psychiatric illness
* Any on-going or pending medical, health or disability related litigation, or current pursuit of disability
* Dementia or cognitive deficits
* A danger to self or others
* Current smoker or smoking within the past 6 months
* Current substance use disorder, including alcohol
* Inability to abstain from over-the-counter anti-inflammatories for the duration of the study (needed for plasma cytokine assessment)
* Unwilling to consent to multiple blood draws
* Unwilling or unable to adhere to all study procedures.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
IL-10 Concentration (pg/mL) | Baseline (pre-OMT intervention), and 5-minutes, 30-minutes, and 60-minutes post-OMT
  Serum IL-10 concentration (pg/mL) will be determined using ELISA assays conducted in triplicate using human ELISA Kits from Millipore Sigma according to manufacturer's directions. Cytokine standards will be used to generate a standard curve, and mean absorbance of experimental samples will be plotted to determine concentration. Data will be synthesized using SoftMax Pro v7.1 and analyzed using Microsoft Excel v2405 and GraphPad v10.2.2.
IL-6 Concentration (pg/mL) | Baseline (pre-OMT intervention), and 5-minutes, 30-minutes, and 60-minutes post-OMT
  Serum IL-6 concentration (pg/mL) will be determined using ELISA assays conducted in triplicate using human ELISA Kits from Millipore Sigma according to manufacturer's directions. Cytokine standards will be used to generate a standard curve, and mean absorbance of experimental samples will be plotted to determine concentration. Data will be synthesized using SoftMax Pro v7.1 and analyzed using Microsoft Excel v2405 and GraphPad v10.2.2.
IL-1β Concentration (pg/mL) | Baseline (pre-OMT intervention), and 5-minutes, 30-minutes, and 60-minutes post-OMT
  Serum IL-1β concentration (pg/mL) will be determined using ELISA assays conducted in triplicate using human ELISA Kits from Millipore Sigma according to manufacturer's directions. Cytokine standards will be used to generate a standard curve, and mean absorbance of experimental samples will be plotted to determine concentration. Data will be synthesized using SoftMax Pro v7.1 and analyzed using Microsoft Excel v2405 and GraphPad v10.2.2.
TNF-α Concentration (pg/mL) | Baseline (pre-OMT intervention), and 5-minutes, 30-minutes, and 60-minutes post-OMT
  Serum TNF-α concentration (pg/mL) will be determined using ELISA assays conducted in triplicate using human ELISA Kits from Millipore Sigma according to manufacturer's directions. Cytokine standards will be used to generate a standard curve, and mean absorbance of experimental samples will be plotted to determine concentration. Data will be synthesized using SoftMax Pro v7.1 and analyzed using Microsoft Excel v2405 and GraphPad v10.2.2.

CONTACTS AND LOCATIONS:
Overall Officials: Kathaleen Briggs Early, PhD, RDN, CDCES, Principal Investigator — PNWU-COM
Locations (1):
- Pacific Northwest University of Health Sciences (PNWU), Yakima, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Investigators have very little data to share from this pilot study. Investigators collected venous blood samples from just 13 people. The study has limited demographic data (age, sex, perceived stress scores), baseline CMP, CBC, and cytokine data.